CLINICAL TRIAL: NCT03961906
Title: Design and Validation of a Modular Physiotherapy Concept for the Treatment of Hereditary Spastic Spinal Paralysis (HSP) - a Randomized Study
Brief Title: Physiotherapy in Hereditary Spastic Paraplegia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ludger Schöls, Principal Investigator, University Hospital Tuebingen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Physiotherapy in HSP
Record Dates: First submitted 2019-05-20; First posted 2019-05-23 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Hereditary Spastic Paraplegia
MeSH Terms: conditions — Spastic Paraplegia, Hereditary | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking only for baseline visit.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tübingen physiotherapy concept (Active Comparator): Will receive our therapy concept and perform self-trainings on a regular basis.
  Interventions: Behavioral: physiotherapy
- controls (No Intervention): Will receive standard-care which includes their regular physiotherapy as provided by the local therapist and can include self-trainings as well.

INTERVENTIONS:
Behavioral: physiotherapy — Will receive two trainings. First training in week one after baseline assessment for three consecutive days 60 min twice daily by trained physiotherapists and in week three further two days with 60min once daily.
  Arms: Tübingen physiotherapy concept

SUMMARY:
Goal of this study is to develop and evaluate a physiotherapy concept that is focused on bilateral leg spasticity and aims to reduce spastic gait disturbance and to improve mobility in patients suffering from HSP.

DETAILED DESCRIPTION:
This is a randomized single-center parallel study with a control group design. A blinded block randomization in groups of four was performed in equal parts toward the treatment (TPC) or the control (regular standard-of-care) group using randomization.com. Group assignment was kept in a closed envelope which was opened by the participant at the end of the baseline visit. Therefore both, the movement disorder specialist as well as the physiotherapist, were blinded to the randomization result for the baseline assessment up to the beginning of the first physiotherapy training session.

Therapeutic effects were evaluated at follow-up visits after 12 weeks (first visit, short-term effect) and after 26 weeks (second visit, long-term effect) comparing standard-of care with the TPC. Clinical evaluation is stated in detail below. Primary outcome assessment of this study was the change between baseline and follow-up assessment in treatment to control group in the spastic paraplegia rating scale (SPRS) score as a validated measure of disease severity (see Reference). Secondary outcome assessment was the change in walking distance in the Three-Minute-Walking test (3MW). Further exploratory outcome assessments were evaluated as effect sizes as specified below.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of hereditary spastic paraplegia
* manifest spastic gait disturbance
* remaining walking ability of at least 100m in three minutes,
* no botulinum toxin treatment during the entire study and three months prior to study inclusion
* no functional electronic stimulation during the study period.

Exclusion Criteria:

* see above

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-03-30 (Actual); Study Completion 2017-03-30 (Actual)

PRIMARY OUTCOMES:
Change in total Spastic paraplegia rating scale (SPRS) score | 12 weeks and 26 weeks
  Change in the total SPRS score (see references for publication) (range 0-52 points, higher points indicated stronger disease severity) will be evaluated at two timepoints compared to baseline (12 weeks as short-term measure and 26 weeks as long-term measure).

SECONDARY OUTCOMES:
Change in Three Minute Walk | 12 weeks and 26 weeks
  Change in walking distance within three minutes will be assessed two timepoints compared to baseline (12 weeks as short-term measure and 26 weeks as long-term measure).

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Tübingen, Center for Neurology, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No
Available upon request

REFERENCES:
- [Background] Schule R, Holland-Letz T, Klimpe S, Kassubek J, Klopstock T, Mall V, Otto S, Winner B, Schols L. The Spastic Paraplegia Rating Scale (SPRS): a reliable and valid measure of disease severity. Neurology. 2006 Aug 8;67(3):430-4. doi: 10.1212/01.wnl.0000228242.53336.90. PMID 16894103